CLINICAL TRIAL: NCT04713540
Title: The Intensive Care Rehabilitation Experiences of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Patients of Pandemic Hospital in Turkey
Brief Title: Rehabilitation in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Caglar Okur, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: intensive care unit
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It was aimed to evaluate the respiratory functions of patients who were hospitalized in intensive care due to Covid-19 and given respiratory rehabilitation, in-bed positioning, and early mobilization, and the time of leaving the intensive care unit.

DETAILED DESCRIPTION:
According to the clinical classification of the World Health Organization, COVID-19; It manifests itself in a wide spectrum, ranging from mild illness, Pneumonia, Severe pneumonia, Acute respiratory distress syndrome (ARDS), to Sepsis and septic shock, resulting in death. In the presence of acute respiratory failure, a decrease in lung compliance leads to increased respiratory work, impaired blood oxygenation, and rapid and superficial breathing patterns. In this case, minimizing inspiratory effort and maximizing the mechanical efficiency of breathing is the most important approach of treatment. In these clinical conditions, the strength of the respiratory muscles may also be reduced.

The challenge of COVID-19 requires a multidisciplinary approach. Rehabilitative intervention should be a part of the treatment pathway from the early stages of the disease. There is an urgent need to build information based on the most effective non-pharmacological measures to ensure the earliest discharge and best recovery after complex COVID-19 infection. Multimodal rehabilitation at all stages of the disease should be part of a holistic medical approach, but there is still no consensus on the timing and type of intervention.

Early physiotherapy in early-onset acute respiratory distress syndrome in the ICU is a critical therapeutic tool to reduce the complications of immobilization in critical diseases such as myopathy, neuropathy and ventilator dependence. Benefits include improved residual respiration, musculoskeletal system, neurological and psychological function; It prevents re-hospitalizations in the medium and long term, improves health status and improves the perceived quality of life after discharge. In an acute setting, interventions can also motivate active recipients to participate in rehabilitation pathways and improve adherence to treatment after discharge.

Serious cases of COVID-19 are associated with the consequences of respiratory support and rehabilitation needs related to prolonged immobility and bed rest. These can include:

Impaired lung function;

* physical impairment and muscle weakness; Delirium and other cognitive disorders; Impaired swallowing and communication; and
* Mental health disorders and psychosocial support needs. Based on this information, we aimed to investigate whether respiratory rehabilitation, positioning, normal joint movement exercises and early mobilization are effective in the treatment of Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Those who have been hospitalized since 11.01.2020
* Those who have been consulted in the physical therapy clinic since 11.01.2020

Exclusion Criteria:

* Fever ˃38.0 °
* Initial consultation time ˂7 days
* Those with ≤3 days from the onset of the disease to shortness of breath
* Chest radiographic scans showing 50% progression within 24 to 48 hours
* With Spo2 level ≤95%
* Resting blood pressure ˂90 / 60 (1mmHg = 0.133kPa) or ˃140 / 90mmHg.

  -˃100 heart rate per minute
* Those with moderate and / or severe heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with covid-19
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Glaskow coma scale | Change from Baseline Glaskow coma scale at 6 months
  The Scale was described in 1974 by Graham Teasdale and Bryan Jennett (Assessment of coma and impaired consciousness. A practical scale. Lancet 1974; 2:81-4.) as a way to communicate about the level of consciousness of patients with an acute brain injury.
APACHE II | Change from Baseline mMRC Dyspnea Scale at 6 months
  APACHE II ("Acute Physiology And Chronic Health Evaluation II") is a severity-of-disease classification system (Knaus et al., 1985),[1] one of several ICU scoring systems. It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
mMRC Dyspnea Scale | Change from Baseline mMRC Dyspnea Scale at 6 months
  The mMRC Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases. Describes baseline dyspnea, but does not accurately quantify response to treatment of chronic obstructive pulmonary disease (COPD).

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Çağlar, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkor Dr. Sadi Konuk Research and Training hospital, Istanbul, Turkey (Türkiye)